CLINICAL TRIAL: NCT03269409
Title: Double Blind, Phase I, Randomized, Parallel Group Study of Hip Decompression Compared to Hip Decompression Supplemented at the Point of Care With Adipose Derived Regenerative Cells for Bilateral Pre-Collapse Femoral Head Osteonecrosis
Brief Title: Use of Adipose Derived Regenerative Cells in Bilateral Femoral Head Osteonecrosis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Logistical delays from device manufacturer due to COVID
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Rafael J. Sierra, M.D., Professor of Orthopedics, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16-003846
Record Dates: First submitted 2017-08-29; First posted 2017-08-31 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Osteonecrosis
MeSH Terms: conditions — Osteonecrosis | interventions — Ringer's Lactate

STUDY DESIGN:
Intervention Model Description: Cytori Celution 800/GP System to process ADRC from lipoaspirate at the point of care.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Hip Decompression with lactated ringers (Sham Comparator): Subjects will receive standard of care hip decompression along with an injection of approximately 5 mls. of lactated ringers.
  Interventions: Other: Lactated Ringers
- Hip Decompression with ADRC (Experimental): Subjects in this arm will have Adipose Derived Regenerative Cells (ADRC)harvested through autologous liposuction and processed outside the body using The Celution 800/GP System (Cytori Therapeutics) before having approximately 5 mls. of ADRCs transplanted into the femoral head after standard of care hip decompression.
  Interventions: Device: The Celution 800/GP System (Cytori Therapeutics); Biological: Adipose Derived Regenerative Cells (ADRC)

INTERVENTIONS:
Other: Lactated Ringers — Approximately 5 mls of lactated ringers will be injected after decompression into the hip that does not receive adipose derived regenerative cells.
  Arms: Hip Decompression with lactated ringers
Device: The Celution 800/GP System (Cytori Therapeutics) — The Celution 800/GP System will be used for the preparation of adipose derived regenerative cells from lipoaspirate. The adipose derived regenerative cells will then be transplanted into the hip, post decompression.
  Arms: Hip Decompression with ADRC
Biological: Adipose Derived Regenerative Cells (ADRC) — Subjects in this arm will have Adipose Derived Regenerative Cells (ADRC)harvested through autologous liposuction and processed outside the body using The Celution 800/GP System (Cytori Therapeutics) before having approximately 5 mls. of ADRCs transplanted into the femoral head after standard of care hip decompression.
  Arms: Hip Decompression with ADRC

SUMMARY:
This randomized clinical trial aims to determine if cells from a patient's own adipose tissue is safe and capable of helping regenerate the femoral head in patients with osteonecrosis. The standard of care is known as hip decompression which simply removes dead tissue from the femoral head and creates a new cavity to be filled in by healthy bone. This trial will use hip decompression in one hip and hip decompression supplemented with adipose derived regenerative cells in patients with osteonecrosis in both of their hips.

DETAILED DESCRIPTION:
Preclinical and clinical data suggest that ADRC may serve as a safe and efficacious adjuvant agent for the treatment of ON. However, to the authors knowledge no RCT in the United States has formally evaluated safety of ADRC in the setting of ON. Therefore, the primary endeavor of this Phase I pilot study will be to evaluate safety of ADRC for pre-collapse ON of the femoral head.

The Celution 800/GP System (Cytori Therapeutics, San Diego, USA) for preparation of ADRC from lipoaspirate is currently being evaluated in FDA approved clinical trials including an orthopedic indication (osteoarthritis). In addition, the device has a CE Mark registration in Europe and Class I approval in Japan. As such, it serves as a known platform that produces a clinical grade product for human use. Other devices on the market process lipoaspirate by either mechanical, washing, or centrifugation methods; however, the remaining components of original adipose tissue are significant and impair the regenerative process. Derivation of relatively pure ADRC has been achieved by few devices and the Cytori Celution 800/GP System is the only one to our knowledge with a sufficient safety and efficacy track record enabling multiple investigational device exemption (IDE) approvals. The reagent used (Celase®) is of a clinical and pharmacologic grade for use in humans. The production of Celase is free of mammalian products.

ELIGIBILITY:
Inclusion Criteria

* Males and females 22-70 years of age.
* No articular surface collapse of the femoral heads as measured by MRI.
* Target disease or condition: Bilateral pre-collapse osteonecrosis of the femoral head.
* Atraumatic osteonecrosis of the femoral head (all other etiologies eligible including corticosteroid and alcohol induced osteonecrosis).
* Ability to safely undergo liposuction that will result in the harvest of a sufficient quantity of adipose tissue (approximately 360 mL). A plastic surgeon evaluation will be performed in order to determine adequate adipose tissue is available for harvest.
* Capacity to provide informed consent
* Ability to comply with protocol
* Normal laboratory values of CBC, CRP, AST, ALT, Bilirubin (total & direct), BUN and Creatinine.

Exclusion Criteria:

* Post traumatic femoral head osteonecrosis.
* Osteonecrosis of the femoral head in stages ≥ IIIA according to the Steinberg classification.
* Asymptomatic osteonecrosis on exam
* Flattening of the femoral head (Steinberg classification Type IV) or articular cartilage collapse at the time of core decompression surgery.
* Septic arthritis, stress fracture, or non-osteonecrosis metabolic bone diseases (e.g., Paget's disease of bone, osteogenesis imperfecta, primary hyperparathyroidism, osteopetrosis, and fibrous dysplasia including monostotic, polyostotic, and McCune-Albright syndrome).
* Skeletal immaturity.
* Known history of HIV, or has active Hepatitis B or active Hepatitis C.
* Disease or medication-related disorder of coagulation (i.e., elevated PTT >13.8 seconds, INR >1.2, or low platelet count <150x109/L). Patients on coumadin, heparin products, and novel oral anticoagulants will be excluded. Antiplatelet medications (e.g. aspirin, clopidogrel) are permitted as long as the aforementioned coagulation labs are within the specified range.
* Patients who have aPTT values greater than or equal to 1.8 times the normal limit.
* Patients who are actively or recently received glycoprotein IIb/IIIa inhibitors (abciximab/ ReoPro, Aggrastat/ tirofiban, eptifibatide/ Integrilin)
* All patients who have inadequate fat deposits (i.e. < 200 ml of lipoaspirate from 3 bilateral sites) will be excluded from the study.
* Lumbar radiculopathy, and/or neurogenic or vascular claudication.
* Active Skin infection at the time of surgery
* Active Local bone infection
* Patients in active treatment for cancer or a blood dyscrasia, or having received chemotherapy, radiotherapy or immunotherapy in past 1 year.
* Participation in another clinical study in the past 30 days or concurrent participation in another clinical trial.
* MRI-incompatible internal devices (pacemakers, aneurysm clips, etc).
* Patients with poorly controlled diabetes mellitus (HbA1C ≥ 8%), peripheral neuropathy, or severe vascular problems.
* Patients receiving treatment with hematopoietic growth factors or antivasculogenesis or anti-angiogenesis treatment (e.g., anti-VEGF).
* Patients requiring bisphosphonate treatment for study duration.
* Pregnant or lactating female patients.
* Prisoners.
* Known starch or gentamycin allergy
* Known amylase deficiency
* Laser- or ultrasound-assisted lipoaspiration technique is used during the lipoaspiration procedure
* An adverse event that meets one or more fat harvest stopping rules has occurred during the lipoaspiration procedure
* Positive gram stain result on ADRC product prior to administration
* If final viable cell count of ADRC product is < 34 million

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2021-06-28 (Actual); Study Completion 2021-06-28 (Actual)

PRIMARY OUTCOMES:
Safety, as measured by the type and number of serious adverse events related to Hip Decompression supplemented with autologous ADRC transplantation compared to Hip Decompression alone. | End of the study (24 months)
  Serious adverse events will only include those that are determined to be related to the transplantation of ADRC and/or Hip Decompression.

SECONDARY OUTCOMES:
In vitro laboratory metrics as measured by flow analysis as well as proliferation and differentiation potential of adipose and bone marrow derived mesenchymal stem cells (MSCs). | Preoperative, Month 12, and Month 24
  These immunophenotypic characterizations will be correlated with MRI imaging data and patient reported outcomes.
Initial signals of efficacy as measured by MRI lesion volume quantification and patient reported outcome metrics. | Preoperative, Month 12, and Month 24
  Preoperative MRI, 1 and 2 year postoperative MRI osteonecrotic lesion volume size compared to quality of life and hip function scores.
  The five subscales include 10 items on pain, 5 items for symptoms (3 symptoms items, 2 stiffness items) 17 items for activities for daily living (ADLs), 4 items for sports and recreations, and 4 items for hip related quality of life.
  Scoring: Each question contains five answer choices ranging from never (score of 0) to extreme (score of 4). A normalized score is calculated for each subscale with 0 indicating extreme symptoms and 100 representing no symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael J Sierra, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials